CLINICAL TRIAL: NCT07203040
Title: Acute Effects of Therapeutic Ultrasound on Passive Cervical Muscle Stiffness and Pain in Adults With Neck Pain: A Randomized Controlled Trial
Brief Title: Acute Effects of Therapeutic Ultrasound on Passive Muscle Stiffness and Pain in Patients With Neck Pain
Acronym: TUS-Neck
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Collaborators: Ataturk University (Other); Amasya University (Other); Bangor University (Other)
Responsible Party: Principal Investigator, esedullah akaras, Assistant Professor & Principal Investigator; Department of Physiotherapy and Rehabilitation, Erzurum Technical University, Erzurum Technical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ETU-EC-2025/123
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Neck Pain
Keywords: Neck Pain; Therapeutic Ultrasound; Muscle Stiffness; Myotonometry
MeSH Terms: conditions — Neck Pain | interventions — Ultrasonic Therapy

STUDY DESIGN:
Intervention Model Description: Single-session, parallel-group, randomized, sham-controlled interventional mode
Who Masked: Participant, Outcomes Assessor
Masking Description: Sham ultrasound matches probe movement and duration; device shows normal indicators but delivers no acoustic output. Outcome measurements are performed by a blinded assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Ultrasound (Active) (Experimental): Single session of continuous therapeutic ultrasound applied to painful/stiff cervical musculature (e.g., upper trapezius and suboccipital/cervical extensors) during one clinic visit.
  Interventions: Device: Therapeutic Ultrasound
- Sham Ultrasound (Sham Comparator): Single session mimicking the active procedure (identical probe movement, contact time, and instructions) but without acoustic output.
  Interventions: Device: Sham Ultrasound

INTERVENTIONS:
Device: Therapeutic Ultrasound — Continuous ultrasound applied to painful/stiff cervical muscles during a single clinic visit; frequency 1-3 MHz, intensity 1.0-1.5 W/cm²
  Arms: Therapeutic Ultrasound (Active)
Device: Sham Ultrasound — Single session mimicking active procedure; device displays appear normal but acoustic output is 0 W/cm²; ~10 minutes;
  Arms: Sham Ultrasound

SUMMARY:
This study will test whether one session of therapeutic ultrasound can immediately reduce muscle stiffness and pain in adults with neck pain. Participants aged 18-50 years who report neck pain of at least 3 out of 10 will be randomly assigned to one of two groups: (1) active ultrasound or (2) sham ultrasound. Both groups will receive the same 10-minute procedure with the probe moved slowly over the painful neck muscles; however, the sham device will not deliver ultrasound energy. Before and right after the session, we will measure passive muscle stiffness at standard points on the neck and shoulder muscles using a handheld device and will record pain intensity on a 0-10 scale. We will also record the Neck Disability Index on the same day. The main question is whether active ultrasound produces a larger immediate decrease in muscle stiffness than sham. We will also examine changes in pain and neck function. The session is performed by trained physiotherapists in a clinic setting. Potential risks are minimal (such as temporary warmth or mild skin redness). There is no cost to participate. Results may help guide safe, non-drug treatment options for neck pain.

DETAILED DESCRIPTION:
Background and Rationale. Therapeutic ultrasound is commonly used to manage musculoskeletal pain and stiffness, yet immediate, objective effects on cervical muscle stiffness are not well established. This trial evaluates whether a single session of continuous ultrasound produces a greater immediate reduction in passive cervical muscle stiffness and pain than a sham procedure.

Study Design. Single-session, parallel-group, randomized, sham-controlled clinical trial (1:1). Masking: participants and outcomes assessor (double-blind). Primary purpose: treatment. Setting: outpatient physiotherapy clinics at Erzurum (university/affiliated hospital).

Participants. Adults 18-50 years with neck pain and baseline pain ≥3/10 on a 0-10 scale. Key exclusions include neurological signs suggesting radiculopathy, pregnancy, pacemaker, open skin lesions/infection at the treatment area, and invasive neck treatment within the past 6 weeks.

Interventions.

Active ultrasound: Continuous therapeutic ultrasound applied to painful/stiff cervical musculature (e.g., upper trapezius and suboccipital/cervical extensors) for ~10 minutes. Frequency 1-3 MHz; intensity 1.0-1.5 W/cm² (adjusted to tolerance); slow, overlapping circular probe movement with standard coupling gel.

Sham ultrasound: Identical device appearance, probe movement, contact time, and instructions, but no acoustic output.

Outcomes and Timing.

Primary outcome: Change in passive muscle stiffness (N/m) measured with a handheld myotonometer at predefined points (e.g., sternocleidomastoid, upper/middle/lower trapezius, cervical extensors), averaged over three taps per site.

Secondary outcomes: Pain intensity (0-10) and Neck Disability Index (0-50). All measures are collected immediately before and immediately after the single treatment session during the same clinic visit.

Randomization and Allocation Concealment. A computer-generated sequence with variable block sizes will assign participants 1:1 to active or sham. Group assignments are concealed in sequentially numbered, opaque envelopes (or via a secure electronic system) opened immediately before treatment by a therapist not involved in outcome assessment.

Blinding. Participants are informed that two forms of ultrasound are being compared. The outcomes assessor is blinded to allocation. Therapists delivering the intervention do not perform outcome measurements.

Sample Size. The target sample is 24 participants (12 per group), which is feasible for a single-session, mechanistic trial and expected to detect a moderate to large between-group difference in immediate stiffness change for planning larger studies.

Statistical Analysis. Analyses will follow the intention-to-treat principle. The primary analysis compares pre-to-post change in stiffness between groups using an analysis of covariance (ANCOVA) with baseline stiffness as a covariate. Secondary outcomes are analyzed similarly. Effect sizes and 95% confidence intervals will be reported. Missing post values (if any) will be handled with appropriate single-visit imputation (e.g., baseline-carried-forward sensitivity analysis).

Safety Monitoring. Ultrasound settings follow standard safety guidelines. Expected minor, transient events include warmth or mild skin redness. Adverse events are recorded throughout the visit; any unexpected event stops the session and triggers medical review.

Data Management. Paper/electronic case report forms are stored in locked/secured systems; records are coded with unique IDs. Only authorized personnel have access. Data are retained per institutional policy.

Participant Timeline. Screening and consent → baseline assessments → randomization → one treatment session (~10 minutes) → immediate post-treatment assessments → discharge and adverse-event check.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years

Neck pain with baseline intensity ≥ 3/10 on a 0-10 scale

Able to understand the study procedures and provide written informed consent

No invasive neck treatment within the past 6 weeks

Exclusion Criteria:

* Neurological signs suggesting cervical radiculopathy or serious spinal pathology

Open wounds, infection, or severe skin disease at the treatment area

Pregnancy or implanted pacemaker

Acute cervical trauma or fracture history

Use of other neck-targeted physical therapies or analgesic procedures on the day of assessment

Any condition judged by the investigators to interfere with safe ultrasound application or outcome measurements

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2025-11-25 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in passive cervical muscle stiffness | Baseline (pre-treatment) to immediately after the single 20-minute session (same visit)
  Dynamic stiffness (N/m) recorded with a handheld myotonometer at predefined points (sternocleidomastoid; upper/middle/lower trapezius; cervical extensors). Each site measured 3 taps and averaged; the limb-side with greater baseline pain is prioritized. Higher values indicate greater stiffness. Primary analysis compares between-group difference in change scores, adjusted for baseline.

SECONDARY OUTCOMES:
Change in Neck Disability Index | Baseline to immediately after the session (same visit)
  Total NDI score (0-50); higher scores indicate greater disability. Same-day administration pre- and post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum Technical University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We may share a de-identified dataset and data dictionary after primary analyses are completed and results are published. The decision will depend on journal/publisher policies, institutional guidance, and data protection considerations.